CLINICAL TRIAL: NCT04608292
Title: Quantitative Measurement of Intracranial Interstitial Fluid Flow Using Magnetic Resonance Spectroscopy
Brief Title: Measuring Fluid Flow in the Brain Using Alcohol and MRI in Healthy Participants
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 023-2020
Record Dates: First submitted 2020-10-23; First posted 2020-10-29 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Diagnostic Technics, Neurological
MeSH Terms: conditions — Neurologic Manifestations | interventions — Magnetic Resonance Imaging; Ethanol; Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: The study will begin with the simplest imaging measurements, and only proceed to longer or more complicated measurements if necessary. Re-breathing apparatus will be used only once the imaging measurement has been decided upon, and blood sampling will be used only on a few subjects to confirm the results. Thus, while there are 9 arms to this trial, it is possible that as few as 3 arms will actually be used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Single-voxel MRS (Active Comparator): MRS
  Interventions: Diagnostic Test: Single-voxel MRS; Other: Alcohol ingestion
- Multi-voxel MRSI (Active Comparator): MRSI
  Interventions: Diagnostic Test: Multi-voxel MRSI; Other: Alcohol ingestion
- Magnetization Transfer Imaging (Active Comparator): MTI
  Interventions: Diagnostic Test: Magnetization Transfer Imaging; Other: Alcohol ingestion
- Single-voxel MRS + ClearMate (Active Comparator): MRS+CM
  Interventions: Diagnostic Test: Single-voxel MRS; Other: Alcohol ingestion; Device: ClearMate
- Multi-voxel MRSI + ClearMate (Active Comparator): MRSI+CM
  Interventions: Diagnostic Test: Multi-voxel MRSI; Other: Alcohol ingestion; Device: ClearMate
- Magnetization Transfer Imaging + ClearMate (Active Comparator): MTI+CM
  Interventions: Diagnostic Test: Magnetization Transfer Imaging; Other: Alcohol ingestion; Device: ClearMate
- Single-voxel MRS + ClearMate + Blood Sampling (Active Comparator): MRS+CM+B
  Interventions: Diagnostic Test: Single-voxel MRS; Other: Alcohol ingestion; Device: ClearMate; Diagnostic Test: Blood sampling
- Multi-voxel MRSI + ClearMate + Blood Sampling (Active Comparator): MRSI+CM+B
  Interventions: Diagnostic Test: Multi-voxel MRSI; Other: Alcohol ingestion; Device: ClearMate; Diagnostic Test: Blood sampling
- Magnetization Transfer Imaging + ClearMate + Blood Sampling (Active Comparator): MTI+CM+B
  Interventions: Diagnostic Test: Magnetization Transfer Imaging; Other: Alcohol ingestion; Device: ClearMate; Diagnostic Test: Blood sampling

INTERVENTIONS:
Diagnostic Test: Single-voxel MRS — Diagnostic test is a single voxel MRS scan
  Arms: Single-voxel MRS; Single-voxel MRS + ClearMate; Single-voxel MRS + ClearMate + Blood Sampling
Diagnostic Test: Multi-voxel MRSI — Diagnostic test is a multi-voxel MRS imaging scan
  Arms: Multi-voxel MRSI; Multi-voxel MRSI + ClearMate; Multi-voxel MRSI + ClearMate + Blood Sampling
Diagnostic Test: Magnetization Transfer Imaging — Diagnostic test is a set of magnetic transfer weighted images
  Arms: Magnetization Transfer Imaging; Magnetization Transfer Imaging + ClearMate; Magnetization Transfer Imaging + ClearMate + Blood Sampling
Other: Alcohol ingestion — Participants will ingest an ethanol-containing beverage of approximately 0.5g/kg of ethanol mixed in 355 mL of a non-caffeinated, sugar-free carbonated drink which must be consumed in 5 minutes
Device: ClearMate — Participants will breathe through the ClearMate, an MR-compatible non-rebreathing circuit which provides oxygen and carbon dioxide that quickly decreases a person's blood alcohol level.
  Arms: Magnetization Transfer Imaging + ClearMate; Magnetization Transfer Imaging + ClearMate + Blood Sampling; Multi-voxel MRSI + ClearMate; Multi-voxel MRSI + ClearMate + Blood Sampling; Single-voxel MRS + ClearMate; Single-voxel MRS + ClearMate + Blood Sampling
Diagnostic Test: Blood sampling — Participants will have a peripheral arterial and peripheral venous line inserted and periodic arterial and venous blood samples will be measured for blood alcohol content.
  Arms: Magnetization Transfer Imaging + ClearMate + Blood Sampling; Multi-voxel MRSI + ClearMate + Blood Sampling; Single-voxel MRS + ClearMate + Blood Sampling

SUMMARY:
Intracranial interstitial fluid (ISF) flow is crucial for adequate clearance of extracellular waste products from the brain parenchyma. Recent demonstrations have shown that a deficiency in flow leads to the accumulation of such waste products in neurodegenerative disorders. Unfortunately, no clinical investigation that gives a quantitative measure of ISF flow exists. Such a test could prove very useful in the clinical setting for multiple neurologic disorders by providing a measure of potential diagnostic importance, as well as yielding a means to monitor response to treatment.

The investigators hypothesize that such an investigation can be developed using magnetic resonance spectroscopy to give a quantitative measure of ISF flow, using spectroscopy of ethanol as a dynamic marker of interstitial fluid. Beneficially, the approach is non-invasive. This pilot project aims to develop this technique with proof of concept in healthy volunteers (males in the age range of 20-75).

This pilot project aims to develop the technique, demonstrating its ability to detect ISF flow and potential differences in rates among healthy volunteers. Success at this stage will give rise to this technique being extended to studies involving individuals with various forms of intracranial pathology for comparison with values seen in healthy individuals, with the ultimate goal of it providing a measure of diagnostic significance in multiple clinical scenarios.

DETAILED DESCRIPTION:
Study hypothesis:

Intracranial interstitial fluid (ISF) flow is crucial for adequate clearance of extracellular waste products from the brain parenchyma. Recent demonstrations have shown that its deficiency leads to their accumulation in neurodegenerative disorders. The hypothesis of this project is MRS and/or MTI can be used to give a quantitative measure of intracranial interstitial fluid flow.

Goals:

The primary goal is to provide a quantitative measure of ISF flow rate through the brain parenchyma. This will be performed by making multiple measurements of the characteristic ethanol peak at different time points with MRS or ethanol-related decreases in water saturation signal in MTI, following its ingestion. This will allow the transit of ethanol, which is equal to the transit of ISF, to be obtained and reported using common transport parameters such as time-to-peak (TTP) and mean transit time (MTT).

Secondary objectives include determining a range of values that may be considered normal ranges for ISF flow rates in healthy individuals. This will be helpful in future experiments when such values will be compared with rates measuring for individuals with various different types of intracranial pathology.

INVESTIGATION STUDY DESIGN:

This pilot project will be experimental with the aim of determining the best quantitative criteria from ethanol MRS or MTI labeling of intracranial ISF flow data to give a reliable clearance metric. To achieve this, the initial proof of concept study will involve 10 healthy male volunteers between the ages of 20-75 undergoing the ethanol-MRS or MTI protocol. This work will be quantitative in nature, since discrete MR signals will be measured and analyzed.

Data Collection Study participants will be required to have fasted a minimum of 6 hours prior to initiating the experiment and refrained from alcohol ingestion for 12 hours. A quick screen will be performed by a research team member of the participant's medications, alcohol consumption, and any neurological conditions prior to moving forward with the examination to verify all volunteers meet all inclusion criteria for the study.

Data will be acquired using either magnetic resonance spectroscopy (MRS), magnetic resonance spectroscopic imaging (MRSI), or magnetization transfer imaging (MTI). A relatively short acquisition (5-7 minutes) will be repeated to acquire a time course for ethanol transit through the brain.

Each study participant will undergo pre-ethanol ingestion MR acquisition. The volunteer will then be given an ethanol-containing beverage. The ethanol content will be approximately 0.5 g/kg, mixed in 355 mL of a non-caffeinated, sugar-free carbonated drink as done previously in other human ethanol MRS experiments (7). The drink must be consumed within 5 minutes and may be provided through clear plastic tubing so the subject does not have to be removed from the scanner. Blood alcohol concentration (BAC) levels for this work are not expected to exceed 0.05%, considered a low level, at the end of the experiment.

After consuming the ethanol-containing beverage, scout images will be acquired again to re-localize the voxels for each subsequent spectral image if study participants need to be placed back in the MR scanner (i.e., did not ingest ethanol through tubing). MRS, MRSI, or MTI will be performed at ~5-7 minutes/spectrum or image, repeating the process continuously for 60-90 minutes. During the scanning, the patient may be asked to breathe through the ClearMate (CM), a specially designed, MR-compatible non-rebreathing circuit that provides oxygen and carbon dioxide that quickly decreases a person's blood alcohol level.

After the final acquisition, the patient will be taken to a supervised area where he/she will remain until blood ethanol levels are registered below 0.05% via a standard breathalyzer test. Once the participant has met this requirement and state that they feel safe to leave the premises, they will be free to go within the recommendations of the study and their participation considered to be complete. Breath sampling will be performed at 30-minute intervals if it is still high.

Finally, since the most accurate way to assess the blood alcohol kinetics is by making comparisons of arterial and venous blood levels, peripheral arterial lines will be inserted (by a Sunnybrook staff anesthesiologist) in a few select study participants. Periodic arterial blood samples from these individuals will be measured for the blood alcohol content and compared with the values for blood samples drawn concurrently from the peripheral intravenous line.

ELIGIBILITY:
Inclusion Criteria:

* Ability to consent, effectively communicate with the investigator, and comply with study protocols
* Low consumer of ethanol (less than 6 drinks per week where a drink is 1 oz of distilled spirits, 6 oz wine, 12 oz beer)

Exclusion Criteria:

* Contraindications to MRI
* History of alcohol or substance abuse
* History of liver pathology
* Currently taking medication such as metronidazole which could induce a disulfiram reaction with ethanol

Ages: 20 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Intracranial Interstitial Fluid Flow Rate | Within 1 week of actual measurement
  The calculated flow rate of intracranial interstitial fluid and its standard deviation

SECONDARY OUTCOMES:
Blood alcohol levels | Within 1 week of blood samples
  Level of alcohol in venous and arterial blood during the examination

CONTACTS AND LOCATIONS:
Overall Officials: Greg J Stanisz, PhD, Principal Investigator — Sunnybrook Research Institute; David Mikulis, MD, Principal Investigator — Krembil Research Institute
Locations (1):
- Sunnybrook Research Institute, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No